CLINICAL TRIAL: NCT06058299
Title: A Phase 2, Partially-blinded, Randomised Trial Assessing the Safety and Efficacy of TBAJ-876 or Bedaquiline, in Combination with Pretomanid and Linezolid in Adult Participants with Newly Diagnosed, Drug-sensitive, Smear-positive Pulmonary Tuberculosis
Brief Title: Phase 2 Trial Assessing TBAJ876 or Bedaquiline, with Pretomanid and Linezolid in Adults with Drug-sensitive Pulmonary Tuberculosis
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Global Alliance for TB Drug Development (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NC-009
Record Dates: First submitted 2023-09-22; First posted 2023-09-28 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Pulmonary TB; Pulmonary Tuberculosis; Drug Sensitive Tuberculosis
Keywords: TBAJ-876; Tuberculosis; pretomanid; bedaquiline; linezolid
MeSH Terms: conditions — Tuberculosis, Pulmonary; Tuberculosis | interventions — TBAJ-876; pretomanid; Linezolid; bedaquiline

STUDY DESIGN:
Intervention Model Description: Participants who meet all of the inclusion criteria and none of the exclusion criteria will be randomised in a 1:1:1:1:1 ratio using an interactive response technology that stratifies based on country and severity of disease (AFB 3+ and/or bilateral cavitation) to 1 of the 5 treatment arms:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: TBAJ-876 and the first 8 weeks of bedaquiline will be blinded. Participants randomized to TBAJ-876 or bedaquiline arms will received active TBAJ-876 (and placebo TBAJ876 to blind the dose) and placebo bedaquiline or placebo TBAJ-876 and active bedaquiline
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- TBAJ876 25 mg (Experimental): TBAJ876 25 mg + pretomanid 200 mg + linezolid 600 mg for 8 weeks followed by HR for 7 to 18 weeks
  Interventions: Drug: TBAJ-876; Drug: Pretomanid; Drug: Linezolid; Drug: HR
- TBAJ876 50 mg (Experimental): TBAJ876 50 mg + pretomanid 200 mg + linezolid 600 mg for 8 weeks followed by HR for 7 to 18 weeks
  Interventions: Drug: TBAJ-876; Drug: Pretomanid; Drug: Linezolid; Drug: HR
- TBAJ876 100 mg (Experimental): TBAJ876 100 mg + pretomanid 200 mg + linezolid 600 mg for 8 weeks followed by HR for 7 to 18 weeks
  Interventions: Drug: TBAJ-876; Drug: Pretomanid; Drug: Linezolid; Drug: HR
- BPaL (Active Comparator): Bedaquiline 200 mg + pretomanid 200 mg + linezolid 600 mg for 8 weeks followed by bedaquiline 100 mg + pretomanid 200 mg + linezolid 600 mg for 18 weeks
  Interventions: Drug: Pretomanid; Drug: Linezolid; Drug: Bedaquiline
- 2HRZE/4HR (Active Comparator): Isoniazid (H) + rifampicin (R) + pyrazinamide (Z), ethambutol (E) for 8 weeks followed by HR for 18 weeks (dose based on participant's weight).
  Interventions: Drug: HRZE; Drug: HR

INTERVENTIONS:
Drug: TBAJ-876 — tablet
  Arms: TBAJ876 100 mg; TBAJ876 25 mg; TBAJ876 50 mg
Drug: Pretomanid — 200 mg
  Other Names: PA-824; Dovprela
  Arms: BPaL; TBAJ876 100 mg; TBAJ876 25 mg; TBAJ876 50 mg
Drug: Linezolid — 600 mg
  Other Names: Zyvox
  Arms: BPaL; TBAJ876 100 mg; TBAJ876 25 mg; TBAJ876 50 mg
Drug: Bedaquiline — 200 mg for 8 weeks followed by 100 mg for 18 weeks
  Other Names: Sirturo; TMC207
  Arms: BPaL
Drug: HRZE — Isoniazid (H) + rifampicin (R) + pyrazinamide (Z) plus ethambutol (E) fixed dose combination tablets dosed by weight
  Arms: 2HRZE/4HR
Drug: HR — Isoniazid (H) + rifampicin (R) fixed dose combination tablets dosed by weight
  Arms: 2HRZE/4HR; TBAJ876 100 mg; TBAJ876 25 mg; TBAJ876 50 mg

SUMMARY:
The goal of this clinical trial is to evaluate 3 dose levels of TBAJ876 for 8 weeks in combination with pretomanid and linezolid, compared to 8 weeks of Isoniazid, rifampicin, pyrazinamide and ethambutol (2HRZE), in adult participants with newly diagnosed, smear-positive, pulmonary drug sensitive tuberculosis (DS-TB).

The main questions the trial aims to answer are:

* What is the optimal dose of TBAJ876 to continue further in development.
* What is the bactericidal activity of bedaquiline with pretomanid and linezolid (B-Pa-L) compared to 2HRZE and TBAJ876-Pa-L over 8 weeks
* What is the efficacy and safety of the 26-week B-Pa-L regimen compared with the SOC (2HRZE/4HR) in participants with DS-TB.

Participants will be seen regularly during treatment (up to 26 weeks) and follow-up (52 weeks post treatment) for safety and efficacy assessments, including but not limited to:

* Safety labs, ECGs, vital signs, physical exams, PK sampling, neuropathy assessments and adverse event monitoring
* Sputum collection

DETAILED DESCRIPTION:
Participants will be treated up to 26 weeks with either:

* TBAJ876 25 mg + pretomanid 200 mg + linezolid 600 mg for 8 weeks followed by HR for 7 to 18 weeks
* TBAJ876 50 mg + pretomanid 200 mg + linezolid 600 mg for 8 weeks followed by HR for 7 to 18 weeks
* TBAJ876 100 mg + pretomanid 200 mg + linezolid 600 mg for 8 weeks followed by HR for 7 to 18 weeks
* Bedaquiline 200 mg + pretomanid 200 mg + linezolid 600 mg for 8 weeks followed by bedaquiline 100 mg + pretomanid 200 mg + linezolid 600 mg for 18 weeks
* Isoniazid (H) + rifampicin (R) + pyrazinamide (Z), ethambutol (E) for 8 weeks followed by HR for 18 weeks (dose based on participant's weight).

TBAJ876 and bedaquiline will be blinded during the first 8 weeks of trial treatment; participants randomised to the TBAJ876 or bedaquiline arms will receive open-label pretomanid and linezolid. Participants randomised to the 2HRZE/4HR arm will receive open-label HRZE.

After receiving 8 weeks of treatment, participants randomised to the TBAJ876-Pa-L treatment arms will receive open-label HR for at least 7 weeks. Treatment completion will be allowed at Week 15 in participants randomised to the TBAJ876-Pa-L arms, if the below criteria are met:

* Week 8 or EOT Make-up Period 1 sputum MGIT culture is negative, and
* The participant has no TB-related symptoms by Week 15. Participants with symptoms that have a more likely alternative explanation are eligible to complete treatment at Week 15.

If the MGIT result is MTB positive and/or there are still TB symptom(s), participants will continue to receive HR (in the 3 TBAJ876 arms) and will complete 18 weeks of treatment with HR, for a total of 26 weeks of treatment. After receiving 8 weeks of trial treatment, all participants randomised to the HRZE arm will receive open-label HR for 18 weeks, for a total of 26 weeks of treatment. After receiving 8 weeks of treatment, a participants randomised to the B-Pa-L arm will receive open-label bedaquiline 100 mg (a reduction from the 200 mg daily dose in the first 8 weeks), pretomanid 200 mg, and linezolid 600 mg daily for 18 weeks, for a total of 26 weeks of trial treatment.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* DS-TB as defined as sensitive to rifampicin and isoniazid by rapid sputum-based test AND either newly diagnosed for TB or have a history of being untreated for at least 3 years after cure from a previous episode of TB
* Of non-childbearing potential OR using effective birth control methods
* Body weight ≥ 35 kg

Exclusion Criteria:

* Karnofsky score < 60 at screening
* Any evidence of extrapulmonary TB
* Cardiovascular or QT prolongation risk factors
* Pregnant or breast-feeding

Any of the following lab toxicities:

* Platelets <100,000/mm³
* Creatinine >1.3 x ULN
* Haemoglobin <9.5 g/dL or <95 g/L
* Absolute neutrophil count <800/mm³
* Serum potassium less than the lower limit of normal for the laboratory.
* ALT and/or AST ≥2.5 x ULN
* Total bilirubin ≥1.6 x ULN
* Direct bilirubin >1 x ULN
* Haemoglobin A1c ≥8.0%
* Total lipase ≥1.5 x ULN
* Total amylase ≥1.5 x ULN
* CPK >3 x ULN (if >3 x ULN, enquire about the participant's recent strenuous activity and consider repeating the test within the screening window)
* TSH >1 x ULN
* Positive results at screening for HBsAg, HAV IgM, or hepatitis C antibodies

For participants living with HIV only:

* CD4+ count<200 cells/μL.
* WHO Clinical Stage 4 HIV disease
* Participant does not agree to use DTG/TFV/3TC during trial if ARV therapy is indicated, and randomised to the TBAJ876 or the B-Pa-L regimen
* If initiation of ARV therapy is indicate, participants who are known to be intolerant, non-responsive to DTG/TFV/3TC or have DTG/TFV/3TC as a contraindication.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 309 (Actual)
Dates: Start 2023-10-24 (Actual); Primary Completion 2024-12-27 (Actual); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Time to stable sputum conversion | Through 8 weeks of treatment
  Time to stable sputum culture conversion to negative status using data from weekly cultures through 8 weeks of treatment.

SECONDARY OUTCOMES:
Favorable Outcome 26 Weeks after End of Treatment | 26 weeks after end of treatment
  Proportion of participants with a favourable outcome at 26 weeks after the end of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Morounfolu Olugbosi, MD, Study Director — TB Alliance
Locations (22):
- National Center for Tuberculosis and Lung Diseases, Tbilisi, Georgia
- Philippines (3):
  - Care Clinical Trial Group Inc., Dasmariñas
  - Tropical Disease Foundation, Makati City
  - Lung Center of the Philippines, Quezon City
- South Africa (13):
  - Setshaba Research Centre, Soshanguve, Gauteng
  - TASK Eden, George, George
  - Madibeng Centre for Research, Brits
  - TASK Brooklyn, Cape Town
  - University of Cape Town Lung Institute (UCTLI), Cape Town
  - Desmond Tutu Health Foundation, Cape Town
  - Enhancing Care Foundation, Durban
  - Synergy Biomed Research Institute (SBRI), East London
  - TB and HIV Investigative Network (THINK), Hillcrest
  - WITS, Clinical HIV Research Unit (CHRU) Themba Lethu Clinic, Helen Joseph Hospital, Johannesburg
  - Perinatal HIV Research Unit (PHRU), Klerksdorp
  - Isango Lethemba TB Research Unit, Port Elizabeth
  - The Aurum Institute, Rustenburg
- Tanzania (3):
  - NIMR-MBEYA Medical Research Center, Mbeya
  - Kilimanjaro Christian Medical Centre, Moshi
  - National Institute for Medical Research (NIMR), Mwanza
- Uganda (2):
  - Case Western Reserve University- Research collaboration Uganda, Kampala
  - Joint Clinical Research Centre (JCRC), Kampala

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Darpo B, Nedelman J, Bruning-Barry R, Hickman D, Kleiman R, Lombardi A, Xue H. Cardiodynamic evaluation of sorfequiline (TBAJ-876): results from a first-in-human study. Antimicrob Agents Chemother. 2026 Jan 30:e0127325. doi: 10.1128/aac.01273-25. Online ahead of print. PMID 41616265
- [Derived] Olugbosi M, Beumont M, Lombard L, Nedelman J, Timm J, Black T, Bruning-Barry R, Hickman D, Lombardi A, Betteridge M, Egizi E, Marcopulos L, Henderson J, Seidel S, Foraida S, Benhayoun M, Sun E. Protocol for a phase 2, partially blinded, randomized trial assessing the safety and efficacy of sorfequiline or bedaquiline in combination with pretomanid and linezolid in adult participants with newly diagnosed, drug-sensitive, smear-positive pulmonary tuberculosis (NC-009). Trials. 2026 Jan 6;27(1):102. doi: 10.1186/s13063-025-09413-5. PMID 41495827
- [Derived] Komm OD, Tyagi S, Garcia A, Almeida D, Chang Y, Li S-Y, Castillo JR, Converse PJ, Black T, Fotouhi N, Nuermberger EL. Contribution of telacebec to novel drug regimens in a murine tuberculosis model. Antimicrob Agents Chemother. 2025 Jan 31;69(1):e0096224. doi: 10.1128/aac.00962-24. Epub 2024 Dec 9. PMID 39651910